CLINICAL TRIAL: NCT07334236
Title: Energy Ramping Versus Fixed Dose ESWL on Stone-Free Rate (Comparative Study)
Brief Title: Energy Ramping Versus Fixed Dose ESWL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: mohammed Abdelhafez (Other)
Responsible Party: Sponsor-Investigator, mohammed Abdelhafez, Urology Resident , sohag hospital university, Sohag University
Organization: Sohag University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Soh-med--25-11-18MS
Record Dates: First submitted 2026-01-03; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Renal Calculi
MeSH Terms: conditions — Kidney Calculi | interventions — Lithotripsy

STUDY DESIGN:
Intervention Model Description: Randomized Parallel Assignment Randomized, two-arm parallel assignment comparing energy-ramping ESWL versus fixed-dose ESWL; participants randomized 1:1. Treatment allocation is stratified by stone size (<10 mm vs ≥10 mm). Primary outcomes assessed at 3 months post-treatment.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fixed-dose ESWL (Active Comparator): * Start therapeutic/high energy (e.g., 80-100% device max) from therapeutic phase.
  * Total shocks: 2000-3000 adjusted by fragmentation progress and tolerance. Log shocks and cumulative energy.
  Interventions: Procedure: Extracorporeal shock wave lithotripsy
- escalating-dose ESWL (Experimental): * Stepwise escalation: increase energy every 500-1000 shocks (example: 20% → 40% → 60% → 80-100%) until therapeutic energy reached.
  * Total shocks: 2000-3000 adjusted by fragmentation progress and tolerance. Log shocks per step and cumulative energy.
  Interventions: Procedure: Extracorporeal shock wave lithotripsy

INTERVENTIONS:
Procedure: Extracorporeal shock wave lithotripsy — Fixed Voltage (experimental): Subjects receive shock wave therapy at a constant energy level (e.g., 20-22 kV) for the entire duration of the session. Standard delivery includes approximately 3,000 shocks at a frequency of 60-90 shocks per minute.
  Voltage Ramping (control): Subjects receive shock wave therapy starting at a low energy level (e.g., 6-10 kV) for an initial "priming" phase of 100-500 shocks. Energy is then escalated in predefined increments (e.g., 1-2 kV every 250-500 shocks) until reaching the target therapeutic voltage.

SUMMARY:
This clinical trial compares two techniques of extracorporeal shock wave lithotripsy (ESWL) - energy ramping versus fixed dose - in adult patients with renal stones. The study aims to evaluate stone-free rates, retreatment needs, and safety outcomes across multiple clinical sites in Egypt.

DETAILED DESCRIPTION:
This multi-center, randomized controlled trial investigates the impact of energy ramping versus fixed-dose ESWL on stone clearance in patients with solitary renal calculi. Participants will be assigned to either a gradually increasing energy protocol or a constant energy protocol using standardized lithotripter settings. The primary outcome is stone-free rate at two weeks post-treatment, assessed via imaging. Secondary outcomes include retreatment rate, pain scores, adverse events, and procedure duration. The study is conducted under IRB approval from Sohag University and follows international ethical standards for human research.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years.
* Radiopaque renal or proximal/mid ureteral stone ≤20 mm.
* eGFR ≥60 mL/min/1.73 m².
* Fit for ESWL.
* Able to give informed consent and complete follow up.

Exclusion Criteria:

* • Pregnancy.

  * Active, untreated UTI.
  * Uncorrected bleeding disorder or anticoagulation that cannot be stopped.
  * Prior ipsilateral renal surgery.
  * Non radio-opaque stone without reliable imaging.
  * Inability to tolerate ESWL or required anesthesia.

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-03 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | 4 weeks
  Proportion of participants achieving complete stone clearance as confirmed by imaging (ultrasound or CT).

SECONDARY OUTCOMES:
Number of ESWL sessions to achieve SFR. | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided